CLINICAL TRIAL: NCT04294368
Title: Targeted Fortification of Donor Breast Milk in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAS6625
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Prematurity; Extreme; Failure to Thrive in Newborn; Growth Retardation; Growth Failure; Infant Nutrition Disorders
Keywords: Human Milk Analyzer; Miris; Target Fortification; Targeted Fortification; Donor Breast Milk
MeSH Terms: conditions — Premature Birth; Failure to Thrive; Infant Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Control group to receive standard fortification of donor breast milk. Experimental group to receive targeted fortification of donor breast milk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): Standard fortification of breast milk
  Interventions: Dietary Supplement: Similac Human Milk Fortifier Extensively Hydrolyzed Protein Concentrated Liquid; Dietary Supplement: Similac Liquid Protein Fortifier; Dietary Supplement: Nestle Microlipid; Dietary Supplement: Medica Nutrition SolCarb; Other: Analysis with Miris (AB) Human Milk Analyzer
- Experimental (Experimental): Targeted fortification of breast milk
  Interventions: Dietary Supplement: Similac Human Milk Fortifier Extensively Hydrolyzed Protein Concentrated Liquid (Targeted Fortification); Dietary Supplement: Similac Liquid Protein Fortifier (Targeted Fortification); Dietary Supplement: Nestle Microlipid (Targeted Fortification); Dietary Supplement: Medica Nutrition SolCarb (Targeted Fortification); Other: Analysis with Miris (AB) Human Milk Analyzer

INTERVENTIONS:
Dietary Supplement: Similac Human Milk Fortifier Extensively Hydrolyzed Protein Concentrated Liquid — The control group will receive mother's breast milk when it is available. Mother's breast milk will be fortified with 4 packets of Similac Human Milk Fortifier (HMF) per 100 mL. When mother's breast milk is not available, participants will be fed donor breast milk with 4 packets of HMF.
  Arms: Control
Dietary Supplement: Similac Liquid Protein Fortifier — For participants in the control group, additional fortification can be added to the milk for patients in this group in response to poor growth, as is standard of care in the NICU. The standard dose is 1 ml per 30 ml of breast milk.
  Arms: Control
Dietary Supplement: Nestle Microlipid — For participants in the control group, additional fortification can be added to the milk for patients in this group in response to poor growth, as is standard of care in the NICU. The standard dose is 1 ml per 30 ml of breast milk.
  Arms: Control
Dietary Supplement: Medica Nutrition SolCarb — For participants in the control group, additional fortification can be added to the milk for patients in this group in response to poor growth, as is standard of care in the NICU.
  Arms: Control
Dietary Supplement: Similac Human Milk Fortifier Extensively Hydrolyzed Protein Concentrated Liquid (Targeted Fortification) — The experimental group will receive mother's breast milk when it is available. Mother's breast milk will be fortified with 4 packets of Similac Human Milk Fortifier (HMF) per 100 mL. When mother's breast milk is not available, participants will be fed donor breast milk with 4 packets of HMF. For participants in the experimental group, the investigators will continue to add fortification. Two packets of HMF per day will be added until goal fortification is reached.
  Arms: Experimental
Dietary Supplement: Similac Liquid Protein Fortifier (Targeted Fortification) — Participants in the experimental group will receive a dose that will vary depending on the base protein content in the donor breast milk for each particular batch of donor breast milk.
  Arms: Experimental
Dietary Supplement: Nestle Microlipid (Targeted Fortification) — Participants in the experimental group will receive a dose that will vary depending on the base fat content in the donor breast milk for each particular batch of donor breast milk
  Arms: Experimental
Dietary Supplement: Medica Nutrition SolCarb (Targeted Fortification) — Participants in the experimental group will receive a dose that will vary depending on the base carbohydrate content in the donor breast milk for each particular batch of donor breast milk
  Arms: Experimental
Other: Analysis with Miris (AB) Human Milk Analyzer — For participants in both the control and the experimental arms, each batch of donor milk will be analyzed using the Miris Human Milk Analyzer. Manufacturer recommendations for milk analysis will be strictly followed.

SUMMARY:
This study is a randomized controlled trial comparing standard fortification of donor breast milk to targeted fortification of donor breast milk in preterm infants. The purpose of the study is to determine if there is a benefit to target fortifying donor breast milk in the preterm population. The investigators hypothesize that infants receiving targeted fortification of donor breast milk will have improved growth compared to infants receiving standard fortification of donor breast milk.

DETAILED DESCRIPTION:
Breast milk is the best food for premature infants due to its ability to protect infants from necrotizing enterocolitis (NEC) and late onset sepsis. When a premature infant's mother's own milk supply is not enough to provide all the milk that her premature infant needs, donated breast milk is the next best option. One of the downsides of donor breast milk is that it often does not contain as much nutrition for the developing infant compared to the milk of a mother of a premature infant. This means a higher likelihood for poor growth in infant receiving mostly donor breast milk compared to mom's own milk. Due to an inability to easily measure the nutritional content of donor breast milk, standard practice has been to assume that the milk has a certain amount of fat, carbohydrates, and protein. Based on these assumptions, a set amount of additional nutritional fortifier is added to both donor and mom's own breast milk prior to it being given to the infant. Studies show that there is often less nutrition in the donor breast milk to start with than assumed. Technology is now available which uses a small volume sample to measure fat, protein, and carbohydrates in human milk, and hence, calculate the calories in the milk. Using this technology, in this study, the investigators will customize the fortification of donor breast milk by first measuring what is in the milk and then adding any additional fortification that is needed to reach the recommended goals for fat, protein, and carbohydrates. The investigators hypothesize that infants receiving this customized milk, so-called "target" fortified donor breast milk, will have better growth than infants receiving the standard amount of fortification added to their donor breast milk.

The study design involves measurement of macronutrient and calorie content of donor breast milk using a point-of-care human milk analyzer (Miris, AB). The individual macronutrient (protein, fat, and carbohydrate) concentrations will be targeted in the intervention group such that the infant will receive protein of 4 g/kg/day, fat of 6.6 g/kg/day, and carbohydrates of 11.6-13.2 g/kg/day. Fortification will be added in a step-wise fashion daily over a 3-4 day period starting when the infant reaches about 80 ml/kg/day in feeding volume. Fortifiers that may be used in this study include: Abbott Similac Human Milk Fortifier Extensively Hydrolyzed Protein Concentrated Liquid, Abbott Liquid Protein, Nestle Microlipid, and Medica Nutrition SolCarb. Participants in the control arm will receive donor milk that is fortified in the standard fashion at this institution; that is, 4 packets of Human Milk Fortifier will be added to 100 ml of donor breast milk. Additional fortification such as liquid protein or microlipid may be added to the donor milk and mom's own milk in response to poor growth for participants in both groups, as is standard of care in this Neonatal Intensive Care Unit (NICU). Patients in both experimental and control groups will always receive mom's own milk first when it is available. Mom's own milk will not be analyzed and will always be fortified in the standard fashion for both groups. The participants will be studied until they reach 34 weeks corrected gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born </= 30 weeks gestational age
* Birth Weight </= 1500 grams

Exclusion Criteria:

* Parents do no consent to donor milk
* Confounders for poor growth such as congenital heart disease, GI diagnoses such as gastroschisis and omphalocele, and or major congenital anomalies
* Grade III or IV intraventricular hemorrhage diagnoses prior to randomization
* Small for gestational age (<3% on Fenton Growth Curve)
* Failure to initiate fortified feeds prior to 3 weeks of life
* Diagnosis of necrotizing entercolitis prior to randomization
* Diagnosis of early onset sepsis confirmed with positive culture

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Up to 11 weeks
  Weight change in g/kg/day, z-score value, and change in z-score from week-to-week
Change in length | Up to 11 weeks
  Length change in cm/kg/day, z-score value, and change in z-score from week-to-week
Head circumference | Up to 11 weeks
  Head circumference change in cm/kg/day, z-score value, and change in z-score from week-to-week

SECONDARY OUTCOMES:
Total Number of Days of Length of Stay in NICU | Up to 1 year
  Today number of days in the NICU.
Rate of Mortality | Up to one year
  Rate of morality during NICU hospitalization.
Number of Feeding Intolerance Events | Up to 34 weeks corrected gestational age
  The number of feeding intolerance events, defined as 1 or more feeds held.
Number of Necrotizing Enterocolitis Events | Up to 1 year of age
  Number of necrotizing enterocolotis events.
Incidence of Bronchopulmonary dysplasia | Up to 1 year of age
  Incidence of supplemental oxygen requirement at 36 weeks corrected gestational age.
Incidence of Retinopathy of prematurity | Up to 1 year of age
  Incidence of retinopathy of prematurity
Percentage of Feeds with Donor Milk and Mother's Milk | Up to 34 weeks corrected gestational age
  Percent of feeds that are donor milk and mom's own milk.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Garland, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center/ New York - Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) may be shared with other researchers at Columbia University Medical Center at the end of the study for the purposes of creating a neurodevelopmental follow-up study that involves following participants in the study until they reach 2 years (corrected post-natal age) in neurodevelopment follow-up clinic. Permission for future contact is included in the consent form for participants in this study. Only participants who consent to future contact will be approached about a neurodevelopmental follow-up study.

REFERENCES:
- [Background] Arslanoglu S, Boquien CY, King C, Lamireau D, Tonetto P, Barnett D, Bertino E, Gaya A, Gebauer C, Grovslien A, Moro GE, Weaver G, Wesolowska AM, Picaud JC. Fortification of Human Milk for Preterm Infants: Update and Recommendations of the European Milk Bank Association (EMBA) Working Group on Human Milk Fortification. Front Pediatr. 2019 Mar 22;7:76. doi: 10.3389/fped.2019.00076. eCollection 2019. PMID 30968003
- [Background] Billard H, Simon L, Desnots E, Sochard A, Boscher C, Riaublanc A, Alexandre-Gouabau MC, Boquien CY. Calibration Adjustment of the Mid-infrared Analyzer for an Accurate Determination of the Macronutrient Composition of Human Milk. J Hum Lact. 2016 Aug;32(3):NP19-27. doi: 10.1177/0890334415588513. Epub 2015 Jun 2. PMID 26037506
- [Background] Fusch C. Avoiding Postnatal Growth Retardation by Individualized Fortification of Breast Milk: Implications for Somatic and Neurodevelopmental Outcomes. Breastfeed Med. 2019 Apr;14(S1):S15-S17. doi: 10.1089/bfm.2019.0031. No abstract available. PMID 30985203
- [Background] Fusch G, Rochow N, Choi A, Fusch S, Poeschl S, Ubah AO, Lee SY, Raja P, Fusch C. Rapid measurement of macronutrients in breast milk: How reliable are infrared milk analyzers? Clin Nutr. 2015 Jun;34(3):465-76. doi: 10.1016/j.clnu.2014.05.005. Epub 2014 May 17. PMID 24912866
- [Background] Gidrewicz DA, Fenton TR. A systematic review and meta-analysis of the nutrient content of preterm and term breast milk. BMC Pediatr. 2014 Aug 30;14:216. doi: 10.1186/1471-2431-14-216. PMID 25174435
- [Background] Horbar JD, Ehrenkranz RA, Badger GJ, Edwards EM, Morrow KA, Soll RF, Buzas JS, Bertino E, Gagliardi L, Bellu R. Weight Growth Velocity and Postnatal Growth Failure in Infants 501 to 1500 Grams: 2000-2013. Pediatrics. 2015 Jul;136(1):e84-92. doi: 10.1542/peds.2015-0129. PMID 26101360
- [Background] John A, Sun R, Maillart L, Schaefer A, Hamilton Spence E, Perrin MT. Macronutrient variability in human milk from donors to a milk bank: Implications for feeding preterm infants. PLoS One. 2019 Jan 25;14(1):e0210610. doi: 10.1371/journal.pone.0210610. eCollection 2019. PMID 30682200
- [Background] Morlacchi L, Mallardi D, Gianni ML, Roggero P, Amato O, Piemontese P, Consonni D, Mosca F. Is targeted fortification of human breast milk an optimal nutrition strategy for preterm infants? An interventional study. J Transl Med. 2016 Jul 1;14(1):195. doi: 10.1186/s12967-016-0957-y. PMID 27370649
- [Background] Montjaux-Regis N, Cristini C, Arnaud C, Glorieux I, Vanpee M, Casper C. Improved growth of preterm infants receiving mother's own raw milk compared with pasteurized donor milk. Acta Paediatr. 2011 Dec;100(12):1548-54. doi: 10.1111/j.1651-2227.2011.02389.x. Epub 2011 Jul 14. PMID 21707744
- [Background] O'Connor DL, Ewaschuk JB, Unger S. Human milk pasteurization: benefits and risks. Curr Opin Clin Nutr Metab Care. 2015 May;18(3):269-75. doi: 10.1097/MCO.0000000000000160. PMID 25769062
- [Background] Quan M, Wang D, Gou L, Sun Z, Ma J, Zhang L, Wang C, Schibler K, Li Z. Individualized Human Milk Fortification to Improve the Growth of Hospitalized Preterm Infants. Nutr Clin Pract. 2020 Aug;35(4):680-688. doi: 10.1002/ncp.10366. Epub 2019 Jul 3. PMID 31268194
- [Background] Rochow N, Fusch G, Choi A, Chessell L, Elliott L, McDonald K, Kuiper E, Purcha M, Turner S, Chan E, Xia MY, Fusch C. Target fortification of breast milk with fat, protein, and carbohydrates for preterm infants. J Pediatr. 2013 Oct;163(4):1001-7. doi: 10.1016/j.jpeds.2013.04.052. Epub 2013 Jun 12. PMID 23769498
- [Background] Zhu M, Yang Z, Ren Y, Duan Y, Gao H, Liu B, Ye W, Wang J, Yin S. Comparison of macronutrient contents in human milk measured using mid-infrared human milk analyser in a field study vs. chemical reference methods. Matern Child Nutr. 2017 Jan;13(1):10.1111/mcn.12248. doi: 10.1111/mcn.12248. Epub 2016 Feb 23. PMID 26914990